Blackfeet Nation IRB – No: 22-03

Date Approved: 01-26-2023

Chair: Frad Hall, EdD

## Vernon Grant, PhD Assistant Research Professor Center for American Indian and Rural Health Equity Montana State University

NCT05314712

Document date: 04-10-23

Blackfeet Nation IRB – No: 22-03 Date Approved: 01-26-2023

Chair: Brad Hall, EdD

## **Consent Form for Sleep Intervention**

**Project Title:** Assessing sleep in Blackfeet families with K-3<sup>rd</sup> grade children.

**Sponsor:** National Institutes of Health; Heart, Lung, and Blood Institute; Center for American Indian and Rural Health Equity

Investigator(s): Vernon Grant, PhD; Research Team (TBD)

**Purpose:** The purpose of this project is to see how a 9-week sleep intervention helps Blackfeet families improve sleep.

**Questions:** If you have any questions about the study please contact Vernon Grant at <a href="mailto:vernong@bfcc.edu">vernong@bfcc.edu</a>. If you have any questions about your rights as a research participant, you may contact the Chair of the Blackfeet Community College Institutional Review Board, Brad Hall at blackfeetnationirb@gmail.com.

What happens during the sleep intervention: Families that sign up for the study will be enrolled in the sleep intervention for 9-weeks. Before the intervention begins, we will ask you and your child to wear a monitor on your wrist for one week so we can collect data on your sleep and physical activity patterns. We will also meet with you and ask you to fill out some surveys and to collect your height and weight. We will do this before and immediately after the intervention and then again at 3 months, so three times all together.

During the sleep intervention, you will be given access to a private Facebook page where we will be providing sleep content. We will also send you text message reminders that may help you to have a better bedtime routine and to help you get more sleep each night. Much of the sleep content we have for you comes directly from Blackfoot elders that were interviewed and a good amount of the content is in the Blackfoot language. We also have a Blackfoot story book and songs that you can use to help create a bedtime routine and get more sleep each night.

**Payment for participation:** You will receive \$150 at each of the three time points when you wear the activity monitor for one week and complete all surveys. At the end of the 9-week sleep intervention, we will have a feed to celebrate with all the families.

**Risks, inconveniences, and discomforts:** Some participants might have some initial discomfort interacting with others on our private Facebook page. Receiving texts may feel inconvenient at times, but it is our hope that the information provided will be helpful to you and your family.

**Benefits:** You may not benefit from taking part in this study. However, potential benefits are learning about strategies that will help you and your family get more sleep each night. Since Blackfoot language is a significant aspect of our sleep intervention content, you may learn new Blackfoot words and utilize them in your home. Overall, we hope that our families obtain an awareness on the importance of nightly sleep.

**Confidentiality:** Research staff will keep confidential research related records and information from this study. If the results of this study are written in a scientific journal or presented at a scientific meeting, information that might identify you, your child, or the community will not be used. Culturally sensitive topics will not be identified or discussed in any publication, presentation, or formal document unless approved by the BNIRB.

Blackfeet Nation IRB – No: 22-03 Date Approved: 01-26-2023 Chair: Brad Hall, EdD

**Voluntary participation/withdrawal:** Your decision to take part in this project is entirely voluntary. You may refuse to take part in the project, or you may withdraw from the study at any time without penalty or loss of benefits to which you are normally entitled.

## **Participant's Statement of Consent**

I have read the above descriptions of this study. I have been informed of the risks and benefits involved, and all my questions have been answered to my satisfaction. Furthermore, I have been assured that any future questions I may have will also be answered by Dr. Grant. I voluntarily agree to take part in this study. I understand that I will receive a copy of this consent form.

| Printed Name of<br>Participant |
|--------------------------------|
| Signature of Participant |
| Date |